CLINICAL TRIAL: NCT04971018
Title: Impact of Transcutaneous Auricular Vagus Nerve Stimulation on Digestive Symptoms in Systemic Sclerosis
Brief Title: Impact of Transcutaneous Auricular Vagus Nerve Stimulation on Digestive Symptoms in Systemic Sclerosis Systemic Sclerosis
Acronym: AVADIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 38RC20.363
Record Dates: First submitted 2021-07-02; First posted 2021-07-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Systemic Sclerosis
Keywords: Transcutaneous auricular vagus nerve stimulation; Digestive symptoms; ta-VNS
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active ta-VNS (Experimental)
  Interventions: Device: Auricular vagus nerve stimulation
- Sham ta-VNS (Placebo Comparator)
  Interventions: Device: Sham Auricular vagus nerve stimulation

INTERVENTIONS:
Device: Auricular vagus nerve stimulation — Patients will have 20-minutes stimulation sessions at home twice a day during 3 months.
  Arms: Active ta-VNS
Device: Sham Auricular vagus nerve stimulation — Patients will have 20-minutes stimulation sessions at home twice a day during 3 months.
  Arms: Sham ta-VNS

SUMMARY:
The purpose of this study is to assess the effect of transcutaneous auricular vagus nerve stimulation (ta-VNS) on gastrointestinal symptoms and quality of life in systemic sclerosis (SSc) patients.

DETAILED DESCRIPTION:
Conduct of study:

Entry into the study: After informed consent, patients will be randomised into two arms (active or sham stimulation). The person responsible for setting the stimulator will make the randomization via an interactive web response system (IWRS). Only this person will have the knowledge of the group allocated to the patient.

Start of ta-VNS sessions according to the 1st modality of stimulation : The patient will perform 2 stimulation sessions per day at home for 3 months. During this period a clinical research associate will contact the patient to verify that he does not encounter any problems with the stimulator. An evaluation visit will be carried out at the end of these three months by a blind physician.

Wash-out period during 1 month.

Start of ta-VNS sessions according to the 2nd modality of stimulation : The patient will perform 2 stimulation sessions per day at home for 3 months. An evaluation visit will be conducted prior to the start of the sessions and another at the end of the sessions.

ELIGIBILITY:
Inclusion Criteria:

* SSc meeting ACR-EULAR (American College of Rheumatology- European League Against Rheumatism) criteria.
* Treatment by proton pump inhibitor (PPI) initiated for at least 3 months.
* Patient's written consent
* Affiliated with social security system

Exclusion Criteria:

* Patients who have previously received central or peripheral neurostimulation treatment regardless of indication.
* People equipped with an active pacemaker in the area of application of the stimulation electrodes.
* People with dermatological disease in the area of application of stimulation electrodes
* People with recent venous or arterial thrombosis (less than one month)
* People with a cochlear implant near the stimulation site
* People followed for proven heart disease
* Person who are protected under the act
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Effect of ta-VNS on Evolution of Gastrointestinal Quality of life. | Evolution of UCLA-SCTC-GIT 2.0 will be assessed from day 0 to Month 3 for the first step. And from the month 4 to month 7 for the second step
  Comparison between the 2 groups of the evolution of the total score University of California, Los Angeles - Scleroderma Clinical Trial Consortium - Gastrointestinal Tract Instrument, version 2.0 ( UCLA-SCTC-GIT 2.0). This score is specific to the SSc, assessing gastrointestinal symptoms and quality of life, validated in French.

SECONDARY OUTCOMES:
Effect of ta-VNS on quality of life. | Evolution of sHAQ will be assessed from day 0 to Month 3 for the first step. And from the month 4 to month 7 for the second step
  Comparison between the 2 groups of the evolution of the Health Assessment Questionnaire for scleroderma (sHAQ)
Effect of ta-VNS on flexibility of the autonomic nervous system | day 0 to Month 3 for the first step. And from the month 4 to month 7 for the second step
  Comparison between the 2 groups of the evolution of heart rate variability (HRV)
Effect of ta-VNS on anxiety and Depression | HADS will be assessed from day 0 to Month 3 for the first step. And from the month 4 to month 7 for the second step
  Comparison between the 2 groups of the Hospital Anxiety and Depression Scale (HADS). HADS score ranges from 0 (better) to 42 (worse).
Effect of ta-VNS on gastric motility | Day 0 to Month 3 for the first step. And from the month 4 to month 7 for the second step
  Comparison between the 2 groups of the frequency of gastric waves assessed with a electrogastrography.
Effect of ta-VNS on digestive symptomatic treatments used | Day 0 to Month 3 for the first step. And from the month 4 to month 7 for the second step
  Comparison between the 2 groups :
  Description of the treatments taken by patients, the evolution of their posology, the frequency of administration.
Effect of ta-VNS on the number and location of digital ulcers. | Day 0 to Month 3 for the first step. And from the month 4 to month 7 for the second step
  Comparison between the 2 groups of the number and location of digital ulcers.
Effect of ta-VNS on Raynaud's Condition Score (RCS) | Day 0 to Month 3 for the first step. And from the month 4 to month 7 for the second step
  Comparison between the 2 groups of the Raynaud's Condition Score (RCS). RCS is a 10 points scale ranging from 0 (better) to 10 (worse).

CONTACTS AND LOCATIONS:
Locations (1):
- vascular medicine department, University hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No